CLINICAL TRIAL: NCT04499911
Title: Efficacy of Neural Prolotherapy in Treatment of Meralgia Paresthetica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Emmanuel Kamal Aziz Saba, Assistant professor, University of Alexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0303901
Record Dates: First submitted 2020-07-25; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Meralgia Paresthetica
Keywords: Meralgia paresthetica; Neural Prolotherapy; lateral femoral cutaneous nerve
MeSH Terms: conditions — Femoral Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neural prolotherapy (Experimental): Neural prolotherapy using isotonic dextrose 5% in water solution (about 5 ml). The isotonic dextrose 5% in water solution (a total volume of about 5 ml). Subcutaneous perineural injection of dextrose (5%) in sterile water was given once. The injection was administered by using the Lyftgot technique of neural prolotherapy on the lateral aspect of the thigh along the tender areas.
  Interventions: Drug: Isotonic dextrose 5% in water solution

INTERVENTIONS:
Drug: Isotonic dextrose 5% in water solution — The isotonic dextrose 5% in water solution (a total volume of about 5 ml). Subcutaneous perineural injection of dextrose (5%) in sterile water was given once. The injection was administered by using the Lyftgot technique of neural prolotherapy on the lateral aspect of the thigh along the tender areas.
  Other Names: Subcutaneous nerual prolotherapy

SUMMARY:
Meralgia paresthetica is an entrapment neuropathy of the lateral femoral cutaneous nerve. Its main manifestation is neuropathic pain on the lateral aspect of the thigh. Neural prolotherapy has shown improvement and relieve of neuropathic pain.

The aim of the current study was to assess the efficacy of neural prolotherapy (subcutaneous perineural injection of dextrose 5% solution) on reliving pain and improvement of function and quality of life in patients with meralgia paresthetica.

DETAILED DESCRIPTION:
Meralgia paresthetica is a mononeuropathy of the lateral femoral cutaneous nerve (i.e. lateral cutaneous nerve of the thigh). It is known as the lateral cutaneous nerve of the thigh neuralgia. It is due to a lot of etiologies. It is characterized by neuropathic pain, tingling, paresthesia and numbness in the anterolateral aspect of the thigh. The symptoms may be provoked or worsened by prolonged standing and walking. Sitting may alleviate the pain because there is reduction of the tension over the nerve, The treatment of meralgia paresthetica is directed towards the improvement of the symptoms which is mainly pain with subsequent improvement of function and quality of life, as well as, treatment of the etiology. The treatment includes conservative and surgical treatment. Conservative treatment consists of non-pharmacologic treatment and pharmacologic treatment. Surgical treatment takes place in case of failure of the conservative treatment. Surgical options consist of neurolysis and neurectomy.

Neural prolotherapy was reported to improve and relieve of neuropathic pain including that of meralgia paresthetica. Neural prolotherapy is the subcutaneous perineural injection of isotonic dextrose (5%) solution especially at the points of fascial penetration of the sensory nerve. It is the site where the sensory nerve reaches the subcutaneous plane. There are scanty studies assessed this issue.

The aim of the current study was to assess the efficacy of neural prolotherapy (subcutaneous perineural injection of dextrose 5% solution) on reliving pain and improvement of function and quality of life in patients with meralgia paresthetica.

ELIGIBILITY:
Inclusion Criteria:

* The patients had clinical evidence of meralgia paresthetica which was based on the following: (i) the presence of pain, paraesthesia and numbness over the anterior and lateral aspect of the thigh; (ii) exacerbation of these symptoms on walking, standing and hip extension; and (iii) meralgia paresthetica was confirmed electrophysiologically by nerve conduction study with or without somatosensory evoked potentials.
* The symptoms needed to be present for at least three months.
* The patients should be unresponsive to conservative treatment. The conservative treatment included lifestyle modification including weight reduction, activity modification (avoid the use of seat belts) and avoidance of tight underwear (tight garments such as jeans, uniforms); non-steroidal anti-inflammatory drugs and anticonvulsants for neuropathic pain; and physiotherapy.

Exclusion Criteria:

* Diabetes mellitus.
* Endocrine disorders.
* Metabolic disorders.
* Systemic rheumatologic disorders.
* Neurological disorders including peripheral neuropathy, lumbar radiculopathy and lumbar plexopathy.
* Coagulopathy.
* Anticoagulant treatment.
* Current skin or soft tissue infection at or near the site of injection.
* Prior local injection of corticosteroid in the past year for meralgia paresthetica.
* Prior neural prolotherapy in the past year for meralgia paresthetica.
* Prior surgery in the affected thigh region.
* Patients presented with a systemic active inflammatory condition or infection.
* Pregnancy.
* Patients refused to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Patient assessment of the overall symptoms of meralgia paresthetica (pain/ burning sensation/paraesthesia) | 4 weeks
  Patient assessment of the overall symptoms of meralgia paresthetica (pain/ burning sensation/paraesthesia) by using visual analogue scale were evaluated collectively by using VAS. It is a 10-cm horizontal scale) which range from 0 (no meralgia paresthetica symptoms), to 10 (severe intolerable symptoms).

SECONDARY OUTCOMES:
Patient assessment of meralgia paresthetica pain | 4 weeks
  Patient assessment of meralgia paresthetica pain was evaluated by using visual analogue scale. It is a 10-cm horizontal scale which range from 0 (no pain), to 10 (severe intolerable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel K Saba, MD, Principal Investigator — Faculty of Medicine, Alexandria University, Alexandria Governorate, Egypt.
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.